CLINICAL TRIAL: NCT06286956
Title: Rectal Tumor Resection Using the UNI-VEC Multichannel Transanal Access Device
Acronym: UNI-VEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vecmedical Spain, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vec-pr-1901
Record Dates: First submitted 2024-02-12; First posted 2024-02-29 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Rectal Polyp; Rectal Polyps; Rectal Lesion; Sessile Colonic Polyp; Pedunculated Colorectal Polyps
Keywords: First-in-human study; Transanal multi channel device; Medical Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treated with UNI-VEC (Experimental)
  Interventions: Device: Treatment of rectal lesions with UNI-VEC

INTERVENTIONS:
Device: Treatment of rectal lesions with UNI-VEC — Polyp resections

SUMMARY:
The aim of the clinical trial is to investigate whether the use of a new multichannel endoscopic transanal access device (named UNI-VEC) is safe and effective in the resection of a rectal polyp or tumor that sits in the distal part of the colon (up to about 20 cm from the anal margin). This is the first study to test the device in humans, after proving its good performance in preclinical development (preclinical development has included functional laboratory tests and an animal trial).

ELIGIBILITY:
Inclusion Criteria:

* All polyps included in the Paris Classification (Polypoid (0-I): Sessile type (Is), Pedunculated type (Ip), Non-polypoid (0-II, III): Raised type (IIa), Flat type (IIb), Depressed type (IIc), Excavated type (III))
* Lesions located from the anal margin to about 20 cm.
* Extent of at least 2 cm² (polyps 2 cm in diameter or areas of ERM or ESD 2 x 2 cm).
* Well or moderately differentiated tumours. T1: Tumours confined to the mucosa (Tis) and submucosa (T1).
* No positive lymph nodes.
* No lymphatic, vascular or perineural invasion.

Exclusion Criteria:

* Are considered vulnerable subjects.
* They suffer from hematological diseases with altered coagulation of their own or pharmacologically induced coagulation disorders (the use of acetylsalicylic acid (ASA) in doses of 150 mg/day is permitted).
* Have rectal lesions that lie above the pectineal line or extend into the anal canal.
* Local or distant metastasis.
* Have a score of more than 2 points on the Wexner faecal incontinence scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Assess that the use of the device meet the established functional requiremnt of allowing the removal of polyps | During the procedure
  The device must allow the removal of polyps with a minimum size of 2 cm (maximum diameter of the removed polyp measured in mm) in the rectum.

SECONDARY OUTCOMES:
Rate of anorectal hemorrhagic events | During the intervention and 1 week after the intervention.
  Anorectal hemorrhagic events for each patinet will be recorded in a table and the number of events will be counted.
Rate of injuries to the anorectal canal and perianal region | During the intervention and 1 week after the intervention.
  The number of injuries to the anorectal canal and perianal region will be recoreded in a table and then the total number of injuries will be counted.
Assessment of anorectal continence | At 7 and 30 days after the procedure. If anorectal incontinence persists at 30 days: follow-up at 2 months. If anorectal incontinence persists: follow-up at 6 months.
  Anorectal continence will be assesed for each Participant with the Wexner Score

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Bercelona
  - Complexo Hospitalario Universitario de A Coruña, A Coruña, Galicia
  - Hospital Quirón-Salud A Coruña, A Coruña, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Complejo Hospitalario Universitario de Vigo, Vigo, Galicia
  - Hospital La Paz, Madrid, Madrid
  - Hospital Universitario Reina Sofía de Murcia, Murcia, Murcia
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Universitario La Fe, Valencia, València

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: A proposal that describes planned analyses must be submitted, and a data sharing agreement must be signed. The documents could be sent by email.

REFERENCES:
- [Background] Noguera Aguilar JF, Gomez Dovigo A, Alonso Aguirre P, Gonzalez Conde B. Endoscopic submucosal dissection transanal hybrid laparoendoscopic robot-assisted. Cir Esp (Engl Ed). 2023 Apr;101(4):291. doi: 10.1016/j.cireng.2022.07.016. Epub 2022 Jul 28. No abstract available. PMID 35908719
- [Background] Noguera Aguilar JF, Gomez Dovigo A, Aguirrezabalaga Gonzalez J, Gonzalez Conde B, Alonso Aguirre P, Martinez Ares D, Sanchez Gonzalez J, Diez Redondo MP, Maseda Diaz O, Torres Garcia MI, Dacal Rivas A, Delgado Rivilla S, Romero Marcos JM, Ramirez Ruiz P, de Maria Pallares P, Alvarez Gallego M, Gomez Besteiro I. Multicenter clinical trial for the resection of rectal polyps using a new laparoendoscopic hybrid transanal access device. Cir Esp (Engl Ed). 2023 Jun;101(6):435-444. doi: 10.1016/j.cireng.2022.12.001. Epub 2022 Dec 21. PMID 36565988